CLINICAL TRIAL: NCT03211169
Title: Comparative Efficacy of Bile Duct Brushings, Cholangioscopy-Directed Biopsies and Pediatric Forceps Biopsies for Obtaining Diagnostic Tissue From Indeterminate Biliary Strictures
Brief Title: Comparison Bile Duct Brushings, Cholangioscopy-Directed Biopsies and Pediatric Forceps Biopsies in Biliary Strictures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate enrollment
Sponsor: Stanford University (Other)
Collaborators: University of Rochester (Other); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Subhas Banerjee, Associate Professor of Medicine, Division of Gastroenterology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 40988
Record Dates: First submitted 2017-06-30; First posted 2017-07-07 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Cholangiocarcinoma; Stricture; Bile Duct
MeSH Terms: conditions — Cholangiocarcinoma; Constriction, Pathologic

STUDY DESIGN:
Intervention Model Description: Randomized prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pediatric Biopsy Forceps directed biopsies (Experimental): Biopsies of the stricture will be taken with Pediatric Biopsy Forceps after bile duct brushings have been obtained.
  Interventions: Procedure: Biopsies of bile duct stricture with pediatric biopsy forceps
- Cholangioscopy-directed biopsies (Active Comparator): Biopsies of the stricture will be taken under cholangioscopic guidance after bile duct brushings have been obtained.
  Interventions: Procedure: Biopsies of bile duct stricture with cholangioscopy-directed biopsies

INTERVENTIONS:
Procedure: Biopsies of bile duct stricture with pediatric biopsy forceps — Biopsies of the stricture will be taken to evaluate diagnostic yield of Pediatric Biopsy Forceps
  Arms: Pediatric Biopsy Forceps directed biopsies
Procedure: Biopsies of bile duct stricture with cholangioscopy-directed biopsies — Biopsies of the stricture will be taken to evaluate diagnostic yield of cholangioscopy-directed biopsies
  Arms: Cholangioscopy-directed biopsies

SUMMARY:
Prospective, randomized, multi-center study. Investigators will compare diagnostic yield of bile duct brushings, pediatric biopsy forceps biopsies and cholangioscopy-directed biopsies for obtaining diagnostic tissue from biliary strictures.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with obstructive jaundice, and imaging (CT or MRI) suggestive of biliary stricture, without obvious pancreatic mass
2. All patients with obstructive jaundice, and index ERCP suggestive of biliary stricture, without obvious pancreatic mass
3. All patients with obstructive jaundice, and prior ERCP suggestive of biliary stricture
4. Expected patient survival of at least 90 days
5. High likelihood of patient follow-up
6. Patient is able to give a written informed consent
7. Patient is willing and able to comply with the study procedures

Exclusion Criteria:

1. Patients with imaging suggestive of pancreatic tumor
2. Children < 18 years of age
3. Pregnant women
4. Patients with impaired decision-making
5. Healthy volunteers
6. Primary Sclerosing Cholangitis (PSC)
7. Patients with untreated coagulopathy at the time of procedure or ongoing need for anti-coagulation
8. Patients with any contraindication to endoscopic procedure
9. Participation in another investigational study that may directly or indirectly affect the results of this study within 30 days prior to the initial visit
10. Patients unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-07-29 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic tissue obtained as assessed by histologic evaluation of biopsy specimen | 1 week
  Malignancy or no malignancy diagnosis obtained from stricture biopsy

SECONDARY OUTCOMES:
Cost | 2 years
  Cumulative $ from devices used and facility fees with each approach
Radiation Exposure | 2 years
  Total Dose, Fluoroscopy Time, Dose Area Product, Effective dose per fluoroscopy machine readings
Procedure Duration | 2 years
  in minutes
Latency to diagnosis | 2 years
  Duration in days from initial procedure to diagnosis of benign or malignant stricture
Adverse Events | 2 weeks
  (Pancreatitis, Bleeding, Infection, Perforation, Death to be assessed one day, one week post-procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University Medical Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No